CLINICAL TRIAL: NCT04036877
Title: Evaluation of Mood Disorders in Bladder Cancer Patients and Their Primary Caregivers
Brief Title: Mood Disorders Bladder Cancer
Status: Completed | Type: Observational
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Principal Investigator, Elizabeth Wulff-Burchfield, MD, Principal Investigator, University of Kansas Medical Center
Other Study IDs: 144280
Record Dates: First submitted 2019-07-22; First posted 2019-07-30 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2024-11

CONDITIONS: Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Mood Disorder Assessment — Assess depression, anxiety, HRQOL, and financial toxicity in both bladder cancer patients and their caregivers via telephone survey

SUMMARY:
This is a cross-sectional study evaluating mood disorders in bladder cancer patients and their caregivers across the bladder cancer trajectory

ELIGIBILITY:
Inclusion Criteria:

* Patients or caregiver of patient with a histologic diagnosis of bladder cancer of the following subtypes, urothelial carcinoma, adenocarcinoma, or squamous cell carcinoma, within 24 months of survey administration and received treatment at the University of Kansas Health System
* ≥ 18 years of age
* Have a patient-designated primary informal/family caregiver
* Able to speak and read English
* Willing and able to provide informed consent
* Functioning telephone number or access to one

Exclusion Criteria:

* Patients or caregivers of patients with metastatic bladder cancer
* Patients who are unable to designate a primary caregiver
* Patients and caregivers who do not both consent to study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients and caregivers of patients with a diagnosis of bladder cancer who have received treatment at the University of Kansas Health System
Sampling Method: Non-Probability Sample
Enrollment: 358 (Actual)
Dates: Start 2019-09-19 (Actual); Primary Completion 2020-01-14 (Actual); Study Completion 2021-08-04 (Actual)

PRIMARY OUTCOMES:
Severity of depression in bladder cancer patients and their caregivers: Patient-Health Questionnaire-9 | Data will be assessed through study completion, on average one year
  Assessed using Patient-Health Questionnaire-9. A standard questionnaire with 9 questions. Score 5-9 is minimal symptoms, 10-14 is minor depression, 15-19 is major depression moderately severe, and 20-27 is severe major depression.
Severity of anxiety in bladder cancer patients and their caregivers: Generalized Anxiety Disorder-7 | Data will be assessed through study completion, on average one year
  Assessed using Generalized Anxiety Disorder-7. A standard questionnaire composed of seven questions with scores ranging from 0 to 21. A score between 5 and 9 indicates mild anxiety, a score between 10 and 14 indicates moderate anxiety, and a score 15 or above indicates severe anxiety.
Health-related quality of life in bladder cancer patients and their caregivers: Short Form-12 | Data will be assessed through study completion, on average one year
  Assessed using Short Form-12. A standard questionnaire with twelve questions, with a score from 0 to 100, where a zero indicates lowest level of health and 100 indicates highest level of health.
Financial Toxicity in bladder cancer patients and their caregivers | Data will be assessed through study completion, on average one year
  Assessed using single-item financial toxicity measure. The measure asks patients to indicate number that best describes their financial stress during pass week from a scale of 0 to 10 with 0 indicating no financial distress and 10 indicating extreme financial distress

OTHER OUTCOMES:
Assess the correlation between caregiver depression, anxiety, and HRQOL and four primary domains of caregiver needs (accessing health services, psychological and emotional needs, work and social needs, and informational needs) | Data will be assessed through study completion, on average one year
  This will be assessed using limited questions from the Supportive Care Needs Survey Partners and Caregivers (SCNS-P&C45) Questionnaire. This questionnaire has one question on health care service needs, two on psychological and emotional needs, three on work and social needs, and two on information needs. Each question is scored from one to five with a higher score indicating higher needs

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Wulff-Burchfield, MD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Health System, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: No